CLINICAL TRIAL: NCT05839964
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Effects of CBN With and Without CBD on Sleep Quality
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Canopy Growth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 710US-1501
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Cannabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CHI-560: Total daily dose: 20 mg CBN (Active Comparator): 2 units (i.e., 2 gummies). Each gummy: 10 mg CBN
  Interventions: Dietary Supplement: CBN and CBD
- CHI-563: Total daily dose: 20 mg CBN + 10 mg CBD (Active Comparator): 2 units (i.e., 2 gummies). Each gummy: 10 mg CBN + 5 mg CBD
  Interventions: Dietary Supplement: CBN and CBD
- CHI-564: Total daily dose: 20 mg CBN + 20 mg CBD (Active Comparator): 2 units (i.e., 2 gummies). Each gummy: 10 mg CBN + 10 mg CBD
  Interventions: Dietary Supplement: CBN and CBD
- CHI-565: Total daily dose: 20 mg CBN + 100 mg CBD (Active Comparator): 2 units (i.e., 2 gummies). Each gummy: 10 mg CBN + 50 mg CBD
  Interventions: Dietary Supplement: CBN and CBD
- CHI-660: Placebo (Placebo Comparator): 2 units (i.e., 2 gummies). Each gummy: Placebo
  Interventions: Dietary Supplement: CBN and CBD

INTERVENTIONS:
Dietary Supplement: CBN and CBD — CBN and CBD in Gummy Format

SUMMARY:
This is a randomized, double-blind, placebo-controlled, study to assess the safety and effects of CHI-560, CHI-563, CHI-564, & CHI-565 versus placebo on sleep quality in healthy adult participants ages 18-55 years.

ELIGIBILITY:
Inclusion Criteria:

1. Person is between 18 and 55-years-old (inclusive).
2. Person has a BMI between 18 and 35 kg/m2 (inclusive).
3. Person is willing and able to provide informed consent.
4. Woman of childbearing potential must not be pregnant or currently breastfeeding.
5. Person agrees to abide by all study restrictions and comply with all study procedures.
6. Person rates past-week sleep quality on a 1 (very poor) to 5 (very good) rating scale as poor (2) or very poor (1).

Exclusion Criteria:

1. Person has a known history of significant allergic condition, significant hypersensitivity to the IP, or allergic reaction to cannabis, cannabinoid medications, hemp products, or excipients of the IP.
2. Person has been exposed to any investigational drug or device < 30 days prior to screening or plans to take an investigational drug in the near future (within 30 days).
3. Person has had a change in allowable medication, caffeine, tobacco, alcohol, supplement, or other drug use dose or regimen within 30 days of screening or has any plans to change dose or regimen during the course of the study.
4. Person has used cannabis, cannabinoid analogue (e.g., dronabinol, nabilone), and/or any CBD- or delta-9-tetrahydrocannabinol (THC)-containing product within 30 days of screening or during the study.
5. Person has history of use of any synthetic cannabinoid receptor agonist (e.g., spice, K2) within the past year.
6. Person is currently using products or medications that may interact with one or more of the ingredients in the IP, including the following drugs or supplements: warfarin, clobazam, valproic acid, phenobarbital, mechanistic target of rapamycin [mTOR] inhibitors, oral tacrolimus, St. John's wort, and Epidiolex.
7. Person has a positive screen (i.e., exceeds cut-point score) for any of the following sleep disorders on the Sleep Disorders Symptom Checklist-17 (SDS-CL-17): narcolepsy, obstructive sleep apnea, restless legs syndrome.
8. Person has a personal or family history (first-degree relative) of a psychotic disorder and/or schizophrenia.
9. Person endorses current suicidal intent as indexed via items 4 and 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS).
10. Person has an acute or progressive disease or disorder that is likely to interfere with the objectives of the study, or the ability to adhere to protocol requirements.
11. Person has a history of cardiovascular disease.
12. Woman of childbearing potential, unless she has not engaged in vaginal intercourse or she has used effective contraception when doing so (for example, oral contraception, double barrier, intra-uterine device) for at least 30 days prior to the study.
13. Woman of childbearing potential, unless willing to ensure that she or her partner use effective contraception (for example, oral contraception, double barrier, intra-uterine device) during the study and for 30 days thereafter (however, a male condom should not be used in conjunction with a female condom).
14. Man whose partner is of childbearing potential, unless willing to ensure that he or his partner use effective contraception (for example, oral contraception, double barrier, intra-uterine device) during the study and for 30 days thereafter (however, a male condom should not be used in conjunction with a female condom).
15. Person has history of diagnosis related to hepatic function and/or significantly impaired hepatic function (alanine aminotransferase [ALT] >5 ⋅ upper limit of normal [ULN] or total bilirubin [TBL] >2 ⋅ ULN) OR the ALT or aspartate aminotransferase (AST) >3 ⋅ ULN and TBL >2 ⋅ ULN (or international normalized ratio [INR] >1.5).
16. Person demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Median sleep quality rating during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning). | Days 1-7
  Median sleep quality rating during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning).

SECONDARY OUTCOMES:
Mean latency to sleep onset during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning). | Days 1-7
  Mean latency to sleep onset during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning).
Number of awakenings after sleep onset during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning). | Days 1-7
  Number of awakenings after sleep onset during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning).
Mean duration of time spent awake after sleep onset during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning). | Days 1-7
  Mean duration of time spent awake after sleep onset during the IP administration phase (measured with the Consensus Sleep Diary - Core Version completed within 1 hour of awakening each morning).
Sleep disturbance during the IP administration phase (measured with the PROMIS completed at the end of the IP administration phase). | Days 1-7
  Sleep disturbance during the IP administration phase (measured with the PROMIS completed at the end of the IP administration phase).
Mean daytime fatigue during the IP administration phase (measured with the VAS-F completed approximately 90 minutes before bedtime each day). | Days 1-7
  Mean daytime fatigue during the IP administration phase (measured with the VAS-F completed approximately 90 minutes before bedtime each day).

OTHER OUTCOMES:
Median early morning awakening rating during the IP administration phase (measured via sleep diary completed within 1 hour of awakening each morning). | Days 1-7
  Median early morning awakening rating during the IP administration phase (measured via sleep diary completed within 1 hour of awakening each morning).
Symptoms of depression during the IP administration phase (measured with the DASS depression subscale completed at the end of the IP administration phase). | Days 1-7
  Symptoms of depression during the IP administration phase (measured with the DASS depression subscale completed at the end of the IP administration phase).
Symptoms of anxiety during the IP administration phase (measured with the DASS anxiety subscale completed at the end of the IP administration phase). | Days 1-7
  Symptoms of anxiety during the IP administration phase (measured with the DASS anxiety subscale completed at the end of the IP administration phase).
Symptoms of general distress during the IP administration phase (measured with the DASS stress subscale completed at the end of the IP administration phase). | Days 1-7
  Symptoms of general distress during the IP administration phase (measured with the DASS stress subscale completed at the end of the IP administration phase).
Irritability during the IP administration phase (measured with the BITe completed at the end of the IP administration phase). | Days 1-7
  Irritability during the IP administration phase (measured with the BITe completed at the end of the IP administration phase).
Perceived psychological stress during the IP administration phase (measured with the PSS completed at the end of the IP administration phase). | Days 1-7
  Perceived psychological stress during the IP administration phase (measured with the PSS completed at the end of the IP administration phase).
Incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs) will be classified by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). | Days 1-7
  Incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs) will be classified by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Feldner, PhD, Principal Investigator — Canopy Growth Corporation
Locations (1):
- Remote, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonn-Miller MO, Feldner MT, Bynion TM, Eglit GML, Brunstetter M, Kalaba M, Zvorsky I, Peters EN, Hennesy M. A double-blind, randomized, placebo-controlled study of the safety and effects of CBN with and without CBD on sleep quality. Exp Clin Psychopharmacol. 2024 Jun;32(3):277-284. doi: 10.1037/pha0000682. Epub 2023 Oct 5. PMID 37796540